CLINICAL TRIAL: NCT03669861
Title: A Prospective, Open-label, Single Center Abatacept in IgG4-Related Disease 10-patient Proof-of-concept Study
Brief Title: Safety and Efficacy of Abatacept in IgG4-Related Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Stone, John H, M.D., M.P.H, Director, Division of Rheumatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-744
Record Dates: First submitted 2018-06-04; First posted 2018-09-13 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: IgG4-related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abatacept (Experimental): To assess the effect of weekly subcutaneous (SC) administration of abatacept on complete remission of IgG4-RD
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Subjects will receive weekly subcutaneous doses of abatacept (125mg) for 24 doses (24 weeks)
  Other Names: Orencia

SUMMARY:
This is a Phase 2, single center, proof of concept clinical trial in subjects with active IgG4-Related Disease (IgG4-RD). Approximately 10 subjects with active IgG4-RD will be enrolled into this study. Subjects will receive weekly subcutaneous doses of abatacept (125mg) for 24 doses (24 weeks).

DETAILED DESCRIPTION:
After obtaining informed consent, all screening procedures and tests establishing eligibility will be performed on the initial screening visit. Subjects determined to be eligible at screening will receive an initial subcutaneous dose of abatacept (125mg), which will be continued weekly for a total of up to 24 doses (24 weeks). Steroid therapy must be tapered off and discontinued over a 4 week period (taper must be completed no later than week 4). Should patients be deemed to have worsening disease or failing therapy at 4 weeks then a trial of steroids can be considered.

Subjects will return on weeks 1, 2, 4, 8, 12, 16, 20, and 24 while on treatment for their injections, and for the scheduled safety and disease response assessments. Subjects will be allowed to self-administer their injections at home. The full treatment period is 24 doses given weekly for 24 weeks. Subjects who are not able to be tapered off corticosteroids or who require reinstitution of corticosteroid therapy at any time during the study will be counted as treatment failures, but may continue on study. Should the IgG4-RD responder index fail to improve by 8 weeks or should there be development of new organ failure at 4 weeks, patient's will be deemed treatment failure and can begin corticosteroid or alternative immunosuppressive therapy at the Investigator's discretion. Those who require rituximab or who require addition of other oral immunosuppressives will be counted as treatment failures and will terminate the study.

All subjects completing the treatment period will have follow up visits off protocolized treatment at 28 and 36 weeks. All adverse events (including serious adverse events (AEs) and deaths) and use of concomitant medication information will be collected throughout the study from screening through study termination. Subjects developing treatment-emergent adverse events or clinically significant safety lab abnormalities will be followed until resolution or until stabilization of the adverse events/abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female 18 years of age or older
2. Meet the American College of Rheumatology (ACR)/EULAR 2018 Classification Criteria for IgG4-RD
3. Have active disease based on an IgG4-RD Responder Index (RI) ≥2 at screening with disease manifestation in at least one organ system excluding lymph nodes at screening
4. May or may not have received prior IgG4-RD therapy
5. Must be willing to taper off any systemic corticosteroid therapy within 4 weeks of first dose of trial drug.
6. Must be able and willing to discontinue any immunosuppressive agent at screening (e.g. methotrexate, mycophenolate mofetil, 6-mercaptopurine, tacrolimus, cyclophosphamide or azathioprine).
7. No history of severe allergic reactions to monoclonal antibodies.
8. Are able and willing to complete the entire study according to the study schedule.
9. Are willing to forego other forms of experimental treatment during the study.
10. Are able to provide written informed consent.

Exclusion Criteria:

1. History or evidence of a clinically unstable/uncontrolled disorder, condition or disease (including but not limited to cardiopulmonary, oncologic, renal, hepatic, metabolic, hematologic or psychiatric) other than IgG4-RD that, in the opinion of the Investigator, would pose a risk to patient safety or interfere with the study evaluation, procedures or completion.
2. Malignancy within 5 years (except successfully treated in situ cervical cancer, resected squamous cell or basal cell carcinoma of the skin, or prostate cancer with no recurrence ≥3 years following prostatectomy).
3. Liver disease: Acute or chronic non-IgG4-related liver disease deemed sufficiently severe to impair their ability to participate in the trial.
4. Uncontrolled disease: evidence of another uncontrolled condition, including drug and alcohol abuse, which could interfere with participation in the trial according to the protocol.
5. Presence of recurrent or chronic infections, defined as ≥3 infections requiring antimicrobials over the past 6 months prior to screening.
6. Active infection requiring hospitalization or treatment with parenteral antimicrobials within the 30 days prior to randomization.
7. Prior use of rituximab (or other B cell depleting agents) within 6 months of enrollment unless B cells have been demonstrated to have repopulated.
8. Use of any investigational agent within 5 half-lives of the agent (or 6 months if the half-life is unknown) prior to enrollment.
9. White blood cell count < 2.5 x 103/µL.
10. Absolute neutrophil count (ANC) < 1.0 x 103/µL.
11. IgG4-related renal disease with serum creatinine >2.0 mg/dL.
12. Hemoglobin < 10 g/dL.
13. Platelet count < 75 x 109/L.
14. Known positive result for HIV I or II antibody, hepatitis B surface antigen, hepatitis B core antibody or hepatitis C antibody.
15. Has received live vaccines within 4 weeks of enrollment.
16. Inability to communicate reliably with the investigator.
17. Patient is pregnant or breast feeding, or planning to become pregnant while enrolled in the study, up to end of study (EOS) visit.
18. Positive pregnancy test at screening or during the study.
19. Subjects who do not agree to use medically acceptable methods of contraception.
20. Male patient with a pregnant partner who is not willing to use a condom during the treatment and up to end of study (EOS)visit.
21. Known or suspected sensitivity to mammalian cell-derived products or any components of the study drug.
22. History of alcohol and/or substance abuse within 12 months prior to screening.
23. Unable or unwilling to partake in follow-up assessments or required protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Stone, MD, Principal Investigator — Massachusetts General Hospital and Harvard Medical School
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon request - without personal health information - following completion of the analysis. Inquiries should be directed to the Principal Investigator.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Concurrent glucocorticoid treatment was permitted but was required to be discontinued by week 4.
Period: Overall Study
Arm/Group | Abatacept
Started | 10
Completed | 3
Not Completed | 7
Not completed — Disease Flare | 5
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: The primary endpoint is 24 weeks, because this is the duration of time patients were on active treatment. The protocol called for a final study visit at 36 weeks, three months after the patients discontinued their active treatment
Groups:
- Abatacept: To assess the effect of weekly subcutaneous (SC) administration of abatacept on complete remission of IgG4-RD. Abatacept: Subjects will receive weekly subcutaneous doses of abatacept (125mg) for 24 doses (24 weeks). The protocol called for a final study visit at 36 weeks, three months after the patients discontinued their active treatment, primarily for safety
Arm/Group | Abatacept
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 64.8 [40 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline Serum IgG4 [Median (Inter-Quartile Range); unit: units on a scale] | 597 [304 to 913]
Baseline Serum IgE [Median (Inter-Quartile Range); unit: IU] | 480.5 [195 to 802]
Disease activity: IgG4-RD Responder Index score [Mean (Full Range); unit: points range 0-75] — Twenty-five domains are assessed in the IgG4-RD RI. If no disease activity is scored in any domain, then the overall score is 0 points (lowest possible value). Scoring refers to manifestations of disease activity present in the last 28 days
  Scoring:
  0 Normal or resolved
  1. Improved but still present
  2. New / Recurrence while patient is off treatment or unchanged from the previous visit*
  3. Worsened or new disease manifestation despite treatment
  Range of score= 0-75 Total score is 75 points (maximum possible score)
  points range 0-75 | 7.2 [2 to 22]
BAS-Duration of IgG4-RD (months) [Mean (Full Range); unit: months] | 54.4 [2 to 240]
Number of active organs affected [Mean (Full Range); unit: count of number of organs involved] | 3.4 [2 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: Effect of weekly subcutaneous (SC) administration of abatacept on complete remission
Time Frame: 24 weeks
Population: The primary outcome, complete remission at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept
Number analyzed (Participants) | 10
Participants | 3

2. Secondary Outcome: Disease Response
Description: Assess the effect of abatacept on disease response at week 12
Time Frame: 12 weeks
Population: All 10 patients were treated initially with abatacept
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept
Number analyzed (Participants) | 10
Participants | 6

3. Secondary Outcome: Disease Response at Week 24
Description: Percentage of patients achieving disease response at week 24
Time Frame: disease response at 24 weeks
Population: disease response at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept
Number analyzed (Participants) | 10
Participants | 5

4. Secondary Outcome: Disease Remission: Flares Over Time Per Subject
Description: number of disease flares per subject
Time Frame: 24 weeks
Population: Subjects with reported disease flare on treatment. Disease flare was defined as recurrence of disease activity or demonstration of a disease exacerbation such that additional therapy beyond the trial protocol was indicated
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Abatacept
Number analyzed (Participants) | 10
units on a scale | 0.2 [0 to 2]

5. Secondary Outcome: Decline in Serum IgG4 Concentration of Responders
Description: Serum IgG4 measured at baseline and week 24
Time Frame: 24 Weeks
Population: serum IgG4 concentration can be used as a surrogate marker for disease activity
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept
Number analyzed (Participants) | 6
Participants | 3

6. Secondary Outcome: Decline in Serum IgE Concentration of Responders
Description: Serum IgE concentration was measured at baseline and Week 24
Time Frame: 24 weeks
Population: Serum IgE concentrations declined in all 6 patients (100%) who demonstrated a disease response with abatacept
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse Event monitoring (from time of study drug administration) to end of study (visit 10 (week 36) or safety follow up visit, if needed). Ten subjects were enrolled in the study between December 2018 and August 2019. Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug a nd that does not necessarily have a causal relationship with this treatment.
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or causes prolongation of existing hospitalization; results in persistent or significant disability/incapacity/congenital anomaly. All Serious Adverse Events (SAEs) that occur following the subject's written consent to participate in the study through 30 days of discontinuation of dosing must be reported.
Arm/Group | Abatacept
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=10)
Myocardial Infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=10)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Thrombocytopenia is a condition in which you have a low blood platelet count. Platelets (thrombocytes) are colorless blood cells that help blood clot. Platelets stop bleeding by clumping and forming plugs in blood vessel injuries
episcleritis (Eye disorders) | 1 (1) — Episcleritis is inflammation of the tissue lying between the sclera (the tough, white, fiber layer covering the eye) and the conjunctiva (the membrane that lines the eyelid and covers the white of the eye).
abdominal pain (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial also comes with additional limitations, specifically the small number of patients, the lack of a comparator group, and the open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-10-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT03669861/Prot_000.pdf